CLINICAL TRIAL: NCT06853808
Title: Prediction Model for Delayed Extubation of Tracheal Intubation in Patients With Maxillofacial Space Infection After Abscess Incision and Drainage Surgery
Acronym: Prediction mod
Status: Not yet recruiting | Type: Observational
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HenanPPH-whb
Record Dates: First submitted 2025-02-15; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Oral Infection
Keywords: oral infection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- normal group: The patient underwent incision and drainage surgery for an abscess in the maxillofacial space, and the endotracheal tube was removed 24 hours later
- Delay group: The patient did not remove the endotracheal tube 24 hours after undergoing incision and drainage surgery for maxillofacial abscess

SUMMARY:
Retrospective exploration of the risk factors associated with mechanical ventilation and tracheal extubation twenty-four hours after abscess incision and drainage surgery in patients with maxillofacial space infection.

DETAILED DESCRIPTION:
1. Retrospective exploration of the risk factors associated with mechanical ventilation and tracheal extubation after 24 hours of abscess incision and drainage in patients with maxillofacial space infection.
2. Prediction model: Based on the identified risk factors, establish a model to predict the risk of tracheal intubation withdrawal 24 hours after abscess incision and drainage surgery in patients with maxillofacial space infection.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old (actual age of the patient)
* Patients diagnosed with maxillofacial space infection upon admission

Exclusion Criteria:

* Serious errors or omissions in key demographic information and medical records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with oral and maxillofacial space infection
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-02-25 (Estimated); Primary Completion 2025-12-25 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Time for extubation of endotracheal tube after surgery | 24hour
  Did the patient remove the endotracheal tube within 24 hours after undergoing maxillofacial abscess incision and drainage surgery.

CONTACTS AND LOCATIONS:
Overall Officials: jiaqiang zhang, Principal Investigator — Department Director

IPD SHARING:
Plan to Share IPD: No